CLINICAL TRIAL: NCT03482973
Title: Pecto-Intercostal Fascial Block for Postoperative Analgesia After Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Associate Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P000044
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease; Sternal Pain
Keywords: Cardiopulmonary Bypass; Cardiac Surgery; Sternotomy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Bupivacaine (Experimental): 20 cc of 0.25% bupivacaine on each side of the sternum at two time points after surgery and POD1
  Interventions: Drug: Bupivacaine Group
- Interventional Placebo (Placebo Comparator): 20 cc of saline on each side of the sternum at two time points after surgery and POD1
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupivacaine Group — 20cc bupivacaine hydrochloride will be administered on each side at two different time points (immediately post operatively and on day 1).
  Arms: Interventional Bupivacaine
Other: Placebo — 20cc placebo (0.9% NaCl) will be administered on each side at two different time points (immediately post operatively and on day 1).
  Arms: Interventional Placebo

SUMMARY:
The purpose of this study is to determine whether administration of a pecto-intercostal fascial plane block (PIFB) with bupivacaine is a more effective therapy for postoperative analgesia after cardiac surgery as compared to patients who receive a sham block of normal saline.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether administration of a pecto-intercostal fascial plane block (PIFB) with bupivacaine is a more effective therapy for postoperative analgesia after cardiac surgery as compared to patients who receive a sham block of normal saline.

Specific Aim 1: To determine whether or not a PIFB with bupivacaine can reduce postoperative pain after cardiac surgery. This will be assessed through:

(Aim 1A) opioid consumption in the first 48 hours postoperatively (Aim 1B) patient self-reported pain scores during their hospital stay

Specific Aim 2: To estimate the effect size in order to obtain information that can be used to power future research on the use of regional modalities of analgesia for cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria

* Patients 18 years of age or older
* Undergoing cardiac surgery with sternotomy, limited to CABG, CABG+valve surgeries and isolated valve surgeries.

Exclusion Criteria

* Current participation in another interventional study
* Preoperative LVEF < 30%
* Use of mechanical circulatory support
* Emergent procedures
* Aortic surgeries, transplants ventricular assist device insertions, bentall, or grafts
* Minimally invasive cardiac procedures or those with thoracotomy approach
* Patients receiving other modalities of regional anesthesia like intrathecal morphine
* Chronic opioid use for chronic pain conditions with tolerance (total daily dose of an opioid at or more than 30 mg morphine equivalent for more than one month within the past year)
* Current use of TCA, gabapentin, or pregabalin
* Hypersensitivity to bupivacaine
* Women who are pregnant or breastfeeding
* Non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 Participants signed consent and none of the participants was withdrawn prior to randomization.
Period: Overall Study
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Bupivacaine | Interventional Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.78 (8.73) | 65.70 (9.86) | 65.73 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 27 | 34 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 8 | 13 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 32 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Weight [Mean (Standard Deviation); unit: Kg] | 86.53 (18.44) | 85.55 (15.10) | 86.04 (16.75)
Height [Mean (Standard Deviation); unit: cm] | 173.73 (12.08) | 172.02 (9.96) | 172.88 (11.03)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 28.57 (5.10) | 28.92 (4.84) | 28.74 (4.94)
Preoperative comorbidities [Number; unit: participants]
  None | 0 | 5 | 5
  Peripheral vascular disease | 2 | 6 | 8
  Connective tissue disease | 0 | 0 | 0
  Ulcer disease | 2 | 4 | 6
  Mild Liver disease | 0 | 0 | 0
  Diabetes without complications | 7 | 8 | 15
  Diabetes with end organ damage | 4 | 5 | 9
  Hemiplegia | 0 | 0 | 0
  Moderate or severe renal disease | 5 | 6 | 11
  Solid tumor (Non-metastatic) | 7 | 6 | 13
  Solid tumor (Metastatic) | 0 | 2 | 2
  Acquired immunodeficiency syndrome (AIDS) | 1 | 0 | 1
  Chronic pain | 8 | 6 | 14
  Hypertension | 31 | 27 | 58
  Hyperlipidemia | 29 | 23 | 52
  Leukemia | 0 | 0 | 0
  Lymphoma or multiple myeloma | 0 | 0 | 0
  Moderate or severe liver disease | 1 | 0 | 1
  Congestive heart failure | 4 | 4 | 8
  Arrhythmia | 6 | 7 | 13
  Coagulopathy | 0 | 0 | 0
  Hypercoagulability | 1 | 1 | 2
  Obesity | 2 | 2 | 4
  Chronic obstructive pulmonary disease(COPD)/Asthma | 6 | 3 | 9
Surgical characteristics [Count of Participants; unit: Participants]
  Isolated Coronary artery bypass grafting (CABG) | 22 | 26 | 48
  CABG surgery + additional surgery | 3 | 5 | 8
  Valve surgery | 14 | 8 | 22
  Other | 1 | 1 | 2
Past surgical history [Number; unit: participants]
  None | 25 | 23 | 48
  Cardiac surgery | 2 | 3 | 5
  Coronary artery stenting | 9 | 6 | 15
  Vascular surgery | 0 | 4 | 4
  Open abdominal surgery | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Total opioid consumption in the first 48 hours post-operatively, measured as milligram morphine equivalents (MME).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: Milligram Morphine Equivalents (MME)
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Number analyzed (Participants) | 40 | 40
Milligram Morphine Equivalents (MME) | 40.8 (22.4) | 49.1 (26.9)

2. Secondary Outcome: Pain Scores
Description: Patient reported pain scores on a scale from 0-10 until discharge for the index admission. Where the minimum score is 0 and, the maximum score is 10. A score of 0 means no pain and the higher the score, the greater the pain intensity, with a score of 10 means worse imaginable pain. Pain scores recorded at 6-8 hourly intervals every day until discharge or 4 days, computed as an average pain score.
Time Frame: At 6-8 hourly intervals every day until discharge or 4 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Number analyzed (Participants) | 40 | 40
score on a scale | 4.8 (2.7) | 5.1 (2.6)

3. Secondary Outcome: ICU Length of Stay
Description: Total duration of stay in ICU for the index admission
Time Frame: Time of ICU admission until time of discharge to hospital floor; through the hospital stay, an average of 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Number analyzed (Participants) | 40 | 40
days | 1.2 [1.0 to 2.8] | 1.7 [1.0 to 3.2]

4. Secondary Outcome: Hospital Length of Stay
Description: Their stay in the hospital for the index admission
Time Frame: Measured in days admitted in the hospital, an average of 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Number analyzed (Participants) | 40 | 40
days | 8 [7 to 11] | 7.5 [6 to 10]

5. Secondary Outcome: Number of Participants With Complications
Description: This includes infection, hematoma, local anesthetic systemic toxicity directly related to the block or the drug used in the block
Time Frame: 7 days post-op on an average
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Bupivacaine | Interventional Placebo
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events will be assessed daily during the hospital stay for a maximum of 4 postoperative days
Description: Anticipated and unanticipated deaths, serious adverse events, and other adverse events due to any cause, whether related or unrelated to study procedures.
Arm/Group | Interventional Bupivacaine | Interventional Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Bupivacaine (N=40) | Interventional Placebo (N=40)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single-center study with restrictive inclusion may place some limitations on generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03482973/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03482973/Prot_SAP_001.pdf